CLINICAL TRIAL: NCT01417208
Title: Clinical Evaluation of the SNaP Wound Care System in Promoting Healing in Chronic Wounds
Status: Withdrawn | Type: Observational
Why Stopped: The study was terminated by Spiraur (original sponsor). Efforts were made to contact the PI/study team members, but were unsuccessful.
Sponsor: KCI USA, Inc (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Organization: Solventum US LLC (Industry)
Other Study IDs: 011711
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Lower Extremity Diabetic Leg Wounds; Lower Extremity Venous Leg Wounds; Lower Extremity Mixed Aetiology Leg Wounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SNaP® Wound Care System
  Interventions: Device: SNaP® Wound Care System

INTERVENTIONS:
Device: SNaP® Wound Care System — Wound dressing applications using customized system. Dressing applications changes per manufacturer recommendation.

SUMMARY:
The purpose of this study is to evaluate a novel topical negative pressure (TNP) wound therapy device called the SNaP® (Smart Negative Pressure) Wound Care System for the treatment of lower extremity diabetic, venous and mixed aetiology leg wounds.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diabetic foot ulceration, venous ulcer, or mixed aetiology ulcer with a surface area <100 cm2 and <10 cm in widest diameter on lower extremity, but larger than 1 cm2 (venous and mixed aetiology ulcers will be defined by clinical exam of treating physician. Diabetic foot ulcers will be defined by clinical exam of the treating physician and as lower extremity ulcers in patients with a diagnosis of diabetes, but without venous stasis disease).
* Wound present for >30 days.
* Patient has wound in location amenable to creation of airtight seal around wound using TNP dressings.
* Patient is able to comply with study protocol requirements.
* Patient is able to understand and provide written consent.

Exclusion Criteria:

* Patient has evidence of wound infection in the opinion of the physician.
* Patient has a thick eschar that persists after wound debridement.
* Patient has an HbA1C >12%.
* Patient has ulcers due to inflammatory conditions such as pyoderma gangrenosum, rheumatoid arthritis, vasculitis, cryoglobulinaemia, necrobiosis lipoidica, panniculitis, lupus erythematosus, scleroderma, or calcinosis.
* Patient has untreated osteomyelitis.
* Patient has any other condition that, in the opinion of the investigator, makes the patient inappropriate to take part in this study.
* Patient is allergic to the wound care device or occlusive dressing.
* Patient has exposed blood vessels.
* Patient is pregnant or pregnancy is suspected.
* Patient is actively participating in other clinical trials that may interfere with their participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetic foot ulceration, venous or mixed aetiology lower limb ulceration who are receiving out-patient treatment from the Section of Wound Healing, Cardiff University, Wales.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Wound Closure | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Wound Healing, Cardiff, Wales, United Kingdom